CLINICAL TRIAL: NCT01948557
Title: A Cohort Study To Assess The Impact Of A Breastfeeding Counselling And Support Strategy To Promote Exclusive Breastfeeding On Post-Natal Transmission Of HIV In African Women
Brief Title: Vertical Transmission Study
Acronym: VTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: WT063009
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: HIV
Keywords: Breastfeeding; Infants; Mother to child transmission of HIV; Survival
MeSH Terms: conditions — Breast Feeding | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infant feeding counselling and support (Other): All mothers provided with counselling. Subsequent support interventions depended on mothers' selection of feeding practice
  Interventions: Behavioral: Infant feeding counselling and support

INTERVENTIONS:
Behavioral: Infant feeding counselling and support — Counselling of appropriate feeding practices as recommended in WHO/UNICEF/UNAIDS guidelines on HIV and infant feeding. Subsequent intensive, home-based support of exclusive breastfeeding or safe replacement feeding according to mothers' selection of feeding practice. Counselling contacts with mothers varied over time. 1-2 antenatal contacts. After delivery, home visits by infant feeding counsellors 3-4 times in first 2 weeks then every 2 weeks until 6 months.
  Outcome data collected by separate field based team who were blinded to mothers HIV status and infant feeding practice.

SUMMARY:
Short courses of drugs can be given to HIV-infected pregnant women to reduce the chance of HIV infection being passed to her child either during pregnancy or during the labour process. However, children can also become infected by drinking the mother's breastmilk which contains the HIV virus. In many poor, developing countries in Africa, breastfeeding is the normal way of infant feeding and is vitally important because of the protection it gives to children from other diseases such as diarrhoea and malnutrition. Ideally there would be a way to make breastfeeding safer from HIV transmission without losing its other advantages.

A medical study recently suggested that HIV-infected women who exclusively breastfed their children i.e. gave breastmilk but without any water, tea, formula milk or any solid foods did not pass on the virus to their children to the same degree as women who MBF with these other fluids and foods. It is important to confirm whether this observation is in fact true or not. We hypothesize that exclusive breastfeeding by HIV-infected mothers carries a lower risk of HIV transmission than mixed breastfeeding.

We propose to follow 2,100 HIV-infected pregnant women and also some HIV-uninfected women from the time that they book at the clinic until 24 months of age. HIV-infected women who say they intend to breastfeed and all the HIV-uninfected women will be visited at their homes by breastfeeding counsellors both before and after delivery to support exclusive breastfeeding. HIV-infected women who choose not to breastfeed will be helped by clinic staff to safely replace all breastmilk with some other milk. An independent team will visit all mothers at their homes and collect information about the way they feed their children. Blood samples will be collected from the children at different times by a simple heel prick and the blood stored on a piece of filter paper. By testing these samples and comparing with the type of feeding at that time, we will be able to see when a child becomes infected and whether exclusive breastfeeding gives any protection.

DETAILED DESCRIPTION:
Short course antiretroviral regimens such as AZT (Thai regimen), or nevirapine (Uganda HIVNET 012 regimen) given to HIV-infected women in pregnancy can reduce in utero and intrapartum transmission to their child by 40-50%. However, these gains are threatened by the continued transmission of HIV through breast milk of poor HIV-infected women in Africa who have no realistic choice but to breastfeed. A recent study from Durban compared for the first time, Mother-to-child transmission of HIV (MTCT) rates in each of the 3 feeding groups viz. exclusive breastfeeding (EBF), mixed breastfeeding (MBF) and formula feeding. The results of this study showed that at 3 months the MTCT in EBF mothers was similar to that in mothers giving only formula feeds, and the MTCT in EBF mothers was significantly lower than in those MBF (14.6% vs. 24.1%). This suggested that EBF may carry no additional risk of MTCT of HIV1 over formula feeding. A prospective study is required to verify these findings.

We propose a cohort study of HIV-infected mothers and their infants, to examine the risk of post-natal transmission of HIV in relation to infant feeding practices after mothers receive intensive breastfeeding counselling and support to practise EBF until about 6 months of age (the optimal duration for EBF).

The hypothesis being tested is: Exclusive breastfeeding by HIV-infected women carries no additional risk of post-natal transmission of HIV than exclusive formula feeding.

The primary objectives of the study are to determine the effect of infant feeding practices on HIV infection rates of infants at 6 and 22 weeks of age, and secondly to to determine the infant survival rate at 24 months of age according to feeding practices and HIV status.

Secondary objectives are:

i) To determine the HIV infection rate of infants as measured of a sample collected within 72 hours of birth; ii) To determine the HIV transmission incidence attributable to the duration of different feeding practices; iii) To determine the cumulative incidence of vertical transmission in EBF, MBF and EFF infants; iv) To describe risk factors, other than feeding practice, for post-natal transmission of HIV, including maternal and infant morbidity and breast health; v) To assess the determinants of transmission in MBF adjusting for exposure factors e.g. type and age of introduction of other food/milk; vi) To describe the morbidity and growth of infants in relation to feeding practices and HIV status; and vii) To describe adherence rates to EBF following a breastfeeding support intervention.

HIV infected women will be counselled according to the WHO/UNICEF/UNAIDS infant feeding guidelines. All HIV-infected women and a random sub-sample of HIV-uninfected women will be recruited antenatally. Those who choose to breastfeed will be visited frequently at home by a team of breastfeeding counsellors before and after delivery to promote and support EBF. HIV-infected mothers who choose not to breastfeed will be supported in their choice by clinic-based staff. An independent team of field monitors will collect data weekly on feeding practices and morbidity of all infants at home visits. Blood samples will be collected by finger/heel prick and stored on filter paper prior to qualitative and quantitative estimation of HIV viral content to determine the timing of transmission.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women attending antenatal clinics in the Mpukunyoni and Hlabisa Tribal Areas of Hlabisa District or at Kwadabeka clinic or St Mary's hospital, Mariannhilll Hospital who offer consent to participate in the study

Exclusion Criteria:

* Intention to leave Hlabisa District or Kwadabeka community within 3 months of delivery.
* Failure to give consent.
* Less than 16 years of age.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3465 (Actual)
Dates: Start 2001-10; Primary Completion 2005-09 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
HIV infection rates of infants who are Exclusively breastfed, Mixed Breastfed or Exclusive Formula Feeding as determined by HIV RNA PCR analysis of a blood sample at that time | 6 weeks of age
HIV infection rates of infants who are Exclusively breastfed, Mixed Breastfed or Exclusive Formula Feeding as determined by HIV RNA PCR analysis of a blood sample at that time | 22 weeks of age
Infant/child survival | 24 months of age

SECONDARY OUTCOMES:
HIV infection rates of infants as determined by HIV RNA PCR analysis of a blood sample obtained in that time period | Within 72 hours of birth
Difference between intrauterine and intrapartum HIV infection rates in women and neonates receiving NVP as determined by HIV RNA PCR analysis of blood samples collected within 72 hours of birth and at 6 weeks | 72 hours and 6 weeks
HIV infection rates of infants at various time points between 6 and 26 weeks, in relation to the type and duration of infant feeding practices i.e. EBF, MBF and EFF (+/- an initial period of EBF) | 6 weeks of age and 26 weeks of age
HIV infection rates of infants 4 weeks after cessation of EBF as determined by HIV RNA PCR analysis of blood samples collected at that time | 4 weeks post cessation of breastfeeding
Prevalent days of diarrhoea | Weekly from birth to 9 months of age
Prevalent days of respiratory distress | Weekly from birth to 9 months of age
Changes in weight, length and head circumference | From birth to 18 months of age
Maternal morbidity | Monthly until 18 months post partum
Percentage of women who adhere to EBF | Until 6 months post partum

CONTACTS AND LOCATIONS:
Overall Officials: Hoosen M Coovadia, MB, Principal Investigator — University of KwaZulu-Natal, and University of the Witwatersand, South Africa; Marie Louise Newell, PhD, Study Chair — University of KwaZulu-Natal and Institute for Child Health, University College, London
Locations (2):
- South Africa (2):
  - Kwadabeka health centre, Durban, KwaZulu-Natal
  - Africa Centre for Health and Population Studies, Somkele, KwaZulu-Natal

REFERENCES:
- [Background] Bland R, Coovadia H, Coutsoudis A, Rollins N, Newell M. Cohort profile: mamanengane or the Africa centre vertical transmission study. Int J Epidemiol. 2010 Apr;39(2):351-60. doi: 10.1093/ije/dyp165. Epub 2009 Mar 31. No abstract available. PMID 19336438
- [Result] Neveu D, Viljoen J, Bland RM, Nagot N, Danaviah S, Coutsoudis A, Rollins NC, Coovadia HM, Van de Perre P, Newell ML. Cumulative exposure to cell-free HIV in breast milk, rather than feeding pattern per se, identifies postnatally infected infants. Clin Infect Dis. 2011 Mar 15;52(6):819-25. doi: 10.1093/cid/ciq203. PMID 21367736
- [Result] Patel D, Bland R, Coovadia H, Rollins N, Coutsoudis A, Newell ML. Breastfeeding, HIV status and weights in South African children: a comparison of HIV-exposed and unexposed children. AIDS. 2010 Jan 28;24(3):437-45. doi: 10.1097/QAD.0b013e3283345f91. PMID 19915445
- [Result] Becquet R, Bland R, Leroy V, Rollins NC, Ekouevi DK, Coutsoudis A, Dabis F, Coovadia HM, Salamon R, Newell ML. Duration, pattern of breastfeeding and postnatal transmission of HIV: pooled analysis of individual data from West and South African cohorts. PLoS One. 2009 Oct 16;4(10):e7397. doi: 10.1371/journal.pone.0007397. PMID 19834601
- [Result] Rollins NC, Becquet R, Bland RM, Coutsoudis A, Coovadia HM, Newell ML. Infant feeding, HIV transmission and mortality at 18 months: the need for appropriate choices by mothers and prioritization within programmes. AIDS. 2008 Nov 12;22(17):2349-57. doi: 10.1097/QAD.0b013e328312c740. PMID 18981775
- [Result] Desmond C, Bland RM, Boyce G, Coovadia HM, Coutsoudis A, Rollins N, Newell ML. Scaling-up exclusive breastfeeding support programmes: the example of KwaZulu-Natal. PLoS One. 2008 Jun 18;3(6):e2454. doi: 10.1371/journal.pone.0002454. PMID 18560596
- [Result] Bland RM, Little KE, Coovadia HM, Coutsoudis A, Rollins NC, Newell ML. Intervention to promote exclusive breast-feeding for the first 6 months of life in a high HIV prevalence area. AIDS. 2008 Apr 23;22(7):883-91. doi: 10.1097/QAD.0b013e3282f768de. PMID 18427207
- [Result] Lebon A, Bland RM, Rollins NC, Coutsoudis A, Coovadia H, Newell ML. Short communication: CD4 counts of HIV-infected pregnant women and their infected children--implications for PMTCT and treatment programmes. Trop Med Int Health. 2007 Dec;12(12):1472-4. doi: 10.1111/j.1365-3156.2007.01954.x. PMID 18076554
- [Result] Bland RM, Becquet R, Rollins NC, Coutsoudis A, Coovadia HM, Newell ML. Breast health problems are rare in both HIV-infected and HIV-uninfected women who receive counseling and support for breast-feeding in South Africa. Clin Infect Dis. 2007 Dec 1;45(11):1502-10. doi: 10.1086/523320. Epub 2007 Oct 22. PMID 17990235
- [Result] Bland RM, Rollins NC, Coovadia HM, Coutsoudis A, Newell ML. Infant feeding counselling for HIV-infected and uninfected women: appropriateness of choice and practice. Bull World Health Organ. 2007 Apr;85(4):289-96. doi: 10.2471/blt.06.032441. PMID 17546310
- [Result] Coovadia HM, Rollins NC, Bland RM, Little K, Coutsoudis A, Bennish ML, Newell ML. Mother-to-child transmission of HIV-1 infection during exclusive breastfeeding in the first 6 months of life: an intervention cohort study. Lancet. 2007 Mar 31;369(9567):1107-16. doi: 10.1016/S0140-6736(07)60283-9. PMID 17398310
- [Result] Rollins NC, Coovadia HM, Bland RM, Coutsoudis A, Bennish ML, Patel D, Newell ML. Pregnancy outcomes in HIV-infected and uninfected women in rural and urban South Africa. J Acquir Immune Defic Syndr. 2007 Mar 1;44(3):321-8. doi: 10.1097/QAI.0b013e31802ea4b0. PMID 17195768
- [Result] Thairu LN, Pelto GH, Rollins NC, Bland RM, Ntshangase N. Sociocultural influences on infant feeding decisions among HIV-infected women in rural Kwa-Zulu Natal, South Africa. Matern Child Nutr. 2005 Jan;1(1):2-10. doi: 10.1111/j.1740-8709.2004.00001.x. PMID 16881874
- [Result] Shah S, Rollins NC, Bland R; Child Health Group. Breastfeeding knowledge among health workers in rural South Africa. J Trop Pediatr. 2005 Feb;51(1):33-8. doi: 10.1093/tropej/fmh071. Epub 2004 Dec 15. PMID 15601651
- [Result] Bland RM, Rollins NC, Van den Broeck J, Coovadia HM; Child Health Group. The use of non-prescribed medication in the first 3 months of life in rural South Africa. Trop Med Int Health. 2004 Jan;9(1):118-24. doi: 10.1046/j.1365-3156.2003.01148.x. PMID 14728615
- [Result] Rollins NC, Dedicoat M, Danaviah S, Page T, Bishop K, Kleinschmidt I, Coovadia HM, Cassol SA; Child Health Group. Prevalence, incidence, and mother-to-child transmission of HIV-1 in rural South Africa. Lancet. 2002 Aug 3;360(9330):389. doi: 10.1016/s0140-6736(02)09599-5. PMID 12241784
- [Result] Bland RM, Rollins NC, Coutsoudis A, Coovadia HM; Child Health Group. Breastfeeding practices in an area of high HIV prevalence in rural South Africa. Acta Paediatr. 2002;91(6):704-11. doi: 10.1080/080352502760069151. PMID 12162606